CLINICAL TRIAL: NCT02274363
Title: Assessment of Psoriasis Severity in Brazilians Patients With Chronic Plaque-type Psoriasis Attending Outpatient Clinics: a Multicenter, Observational, and Cross-sectional Study (APPISOT)
Brief Title: A Study to Assess the Severity of Psoriasis in Brazilians Participants With Chronic Plaque-type Psoriasis
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100727; CNTO1275PSY0001 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis; Plaque
Keywords: Psoriasis; Plaque; Chronic
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Brazilian Participants with Chronic Plaque-type Psoriasis: Brazilian participants with plaque psoriasis followed up at teaching and non-teaching specialized dermatology centers will be included in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants will not receive any intervention in this study. Participants with chronic plaque type psoriasis will be assessed at a single time point, primarily for severity of plaque-type psoriasis Participants will not be followed over time. Data will be collected from the medical consultation notes, medical records and during interviews.

SUMMARY:
The purpose of this study is to assess the severity of plaque-type psoriasis (common genetically determined, chronic, inflammatory skin disease characterized by rounded erythematous, dry, scaling patches. The lesions have a predilection for nails, scalp, genitalia, extensor surfaces, and the lumbosacral region) in brazilian participants with chronic plaque-type psoriasis.

DETAILED DESCRIPTION:
This is a cross-sectional (studies in which the presence or absence of disease or other health-related variables are determined in each member of the study population or in a representative sample at one particular time), observational (clinical study in which participants may receive diagnostic, therapeutic, or other types of interventions, but the investigator does not assign participants to specific interventions), non-interventional, multicenter study (when more than one hospital or medical school team work on a medical research study). Participants with plaque psoriasis will be followed up at specialized dermatology centers. Participants will undergo assessment at a single time point and all assessments will be conducted on the same day. Information will be collected about disease severity/ socioeconomic variables and demographics; clinical characteristics; treatment (current and past procedures and therapies to treat psoriasis); quality of life; and comorbidities identified after plaque psoriasis was diagnosed. The information will be obtained from the medical records, as requested, and during the medical interviews. The primary objective of this study is to assess the severity of plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed with chronic plaque psoriasis
* Participant is at least 18 years old
* Participant is able to understand and sign the Informed Consent Form

Exclusion Criteria:

* In the opinion of the investigator, the participant is unable or unavailable to complete all study procedures
* Participant suffers from a psychiatric condition or any other clinical condition that might interfere with the ability to understand the study requirements
* Participant refuses consent or is unwilling to supply the required information within the required period
* Participant is taking part in an interventionist clinical trial with an investigational agent (i.e. non-commercialized agent) or in an interventionist clinical trial sponsored by Johnson & Johnson
* Participant is an employee of the investigator or study site and is directly involved in the conduction of this study or other studies conducted by the same investigator at the same site, or is a family member of the employee or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants at least 18 years of age with chronic plaque psoriasis under outpatient follow-up will be included irrespective of disease severity.
Sampling Method: Non-Probability Sample
Enrollment: 1131 (Actual)
Dates: Start 2012-04-10 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

PRIMARY OUTCOMES:
Participant's Psoriasis Severity | At single study visit anytime between 6 to 12 months
  Psoriasis severity will be graded as mild or moderate to severe based on psoriasis area and severity index (PASI) score;combined assessment of lesion severity and area affected into single score. Body will be divided into 4 sections:head, arms, trunk, and legs. For each section, percent (%) area of skin involved was estimated:0=0%, 1=less than (<) 10%, 2=10 to <30%, 3=30 to <50%, 4=50 to <70%, 5=70 to <90%, 6=90 to 100%. Severity will be estimated by clinical signs:erythema,induration,desquamation;scale:0= none to 4=maximum. Final PASI=sum of severity parameters for each section*area score*weight of section (head:0.1,arms:0.2,body:0.3,legs:0.4);total possible score range: 0=no disease to 72=maximal disease or on the dermatology life quality index (DLQI);comprises 10 questions evaluated on a scale from 0 (not at all) to 3 (very much). The total scores may range from 0 to 30, with higher scores indicating a higher level of disability or on body surface area (BSA).

SECONDARY OUTCOMES:
Participant Current Psoriasis Severity | At single study visit anytime between 6 to 12 months
  Psoriasis severity will be graded as mild or moderate to severe based on psoriasis area and severity index (PASI) score or on the dermatology life quality index (DLQI) or on body surface area (BSA). Participants with a score greater than (>) 10 in any of these scales will be reported as moderate to severe psoriasis. Participants with a PASI score less than or equal to (<=) 10 will be reported as mild psoriasis. Assessment should consider the participant's status at inclusion.
Disease Duration | Time from disease diagnosis to inclusion (up to 12 months)
  Disease duration is the time from disease diagnosis to inclusion in the study.
Hospital Anxiety and Depression Scale (HADS) Score | At single study visit anytime between 6 to 12 months
  The HADS has been developed to identify symptoms of anxiety and depression in hospitalized participants and in outpatients. It comprises 14 items, seven to assess anxiety (HADS-A), namely items 1, 3, 5, 7, 9, 11, and 13; and seven to assess depression (HADS-D), namely items 2, 4, 6, 8, 10, 12, and 14. Each item receives a score from 0 to 3 on a Likert Scale. The total score for each scale is obtained by adding the individual scores for each item, with the maximum score 21. The presence or absence of depression and anxiety will be defined, for each respective scale, based on the following cutoff values: HADS (anxiety): 0-8 = no anxiety; >9 = anxiety; HADS (depression): 8-8 = no depression; >9 = depression.
Brief Pain Inventory (BPI) Scale Score | At single study visit anytime between 6 to 12 months
  The presence of pain or discomfort over the past week will be assessed using the BPI. The BPI consists of 9 items related to pain (items 3 to 6) and the impact of pain/discomfort (items 9a to 9g) on general activity, mood, walking ability, work, relations with others, sleep and enjoyment of life. Each item is assessed on an 11-point scale varying from zero (no pain or no impact) to 10 (worst possible pain/worst possible impact). The items cover the dimensions of pain/discomfort severity and impact, and the scores are calculated from the means of each item, and may range from 0 to 10. The higher the score, the worse is the pain/discomfort and the perceived impact.
Health Related Quality of Life (HRQoL) Score | At single study visit anytime between 6 to 12 months
  The HRQoL will be assessed using 36-Item Short-Form Health Survey (SF-36), to assess global HRQoL; and the Dermatology Life Quality Index (DLQI) to assess quality of life specifically related to dermatological conditions. The SF-36 comprises 36 questions divided in 8 domains: physical functioning (10 items), role-physical (4 items), bodily pain (2 items), general health (5 items), vitality (4 items), social functioning (2 items), role-emotional (3 items), mental health (5 items), and a question for comparative assessment of current health status with that of the previous year. The domain-specific scores range from 0 (worst status) to 100 (best status). DLQI comprises 10 questions evaluated on a scale from 0 (not at all) to 3 (very much). The total scores may range from 0 to 30, with higher scores indicating a higher level of disability.
Number of Participants With Alcohol Abuse | At single study visit anytime between 6 to 12 months
  Disorders related to alcohol abuse will be investigated using the cut down, annoyed by criticism, guilty and eye-opener (CAGE) questionnaire. CAGE is a brief questionnaire that comprises four questions to be answered affirmatively or negatively. Two affirmative answers warrant a screening for alcohol abuse or dependence.
Number of Participants With Comorbidities | At single stuy visit anytime between 6 to 12 months
  Comorbidity refers to the presence of co-existing or additional diseases with reference to an initial diagnosis or with reference to the index condition that is the subject of study. Participants with Crohn's disease, systemic arterial hypertension, hyperlipidemia, arthritis, obesity, pruritus/burning sensation, depression, ulcerative colitis, metabolic syndrome, neoplasia, diabetes mellitus, ischemic disease and other cardiovascular disorders will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica
Locations (16):
- Brazil (16):
  - Belém
  - Belo Horizonte
  - Botucatu
  - Brasília
  - Campinas
  - Curitiba
  - Fortaleza
  - Goiânia
  - João Pessoa
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - Santo André
  - São José do Rio Preto
  - São Paulo